CLINICAL TRIAL: NCT00097331
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Dose Ranging Study to Investigate the Efficacy and Safety of Three Months Administration of SB-683699 (150 - 1200mg Twice Daily) in Subjects With Relapsing Multiple Sclerosis
Brief Title: Three Months Treatment With SB683699 In Patients With Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683699/003
Record Dates: First submitted 2004-11-22; First posted 2004-11-23 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis; relapsing; remitting; Relapsing-Remitting MS (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence | interventions — Firategrast

INTERVENTIONS:
Drug: SB683699

SUMMARY:
The study will evaluate the effectiveness and safety of the investigational drug SB683699 in treating patients with relapsing multiple sclerosis (MS), using data from magnetic resonance imaging (MRI) scans as the main measure.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of multiple sclerosis (MS).
* Expanded Disability Status Score 0 - 6.5.
* One or more relapse of MS in previous 12 months.
* Currently not taking any medications for MS (apart from those used to treat symptoms).

Exclusion criteria:

* Patients with significantly abnormal laboratory tests or electrocardiogram (ECG) results.
* Subjects who cannot have MRI scans.
* Women who are pregnant, breast feeding or planning to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2004-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Number of new gadolinium-enhancing lesions on monthly MRI scans

SECONDARY OUTCOMES:
Number of other lesion types on MRI
Number of relapses during treatment
Expanded Disability Status Scale (EDSS) and MS Functional Composite (MSFC)
Circulating lymphocyte and neutrophil counts
Health Outcomes: MSIS-29, Employment status

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Fraiture En Condroz
- GSK Investigational Site, Hamburg, Hamburg, Germany
- Poland (3):
  - GSK Investigational Site, Polanki
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Málaga, Spain